CLINICAL TRIAL: NCT01372579
Title: Phase II Neoadjuvant Trial With Carboplatin and Eribulin Mesylate in Triple Negative Breast Cancer Patients
Brief Title: Carboplatin and Eribulin Mesylate in Triple Negative Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 10B07; NCI-2011-00600 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00045038 (Other: Northwestern University IRB#)
Record Dates: First submitted 2011-06-01; First posted 2011-06-14 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-05

CONDITIONS: Estrogen Receptor-negative Breast Cancer; HER2-negative Breast Cancer; Male Breast Cancer; Progesterone Receptor-negative Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — eribulin; Carboplatin; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (neoadjuvant chemotherapy) (Experimental): Patients receive eribulin mesylate IV over 2-5 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: eribulin mesylate; Drug: carboplatin; Procedure: biopsy

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: Halaven; B1939; E7389; ER-086526; halichrondrin B analog
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Procedure: biopsy — Correlative studies
  Other Names: biopsies

SUMMARY:
This phase II trial studies how well giving eribulin mesylate and carboplatin together before surgery works in treating patients with stage I-III triple-negative breast cancer. Drugs used in chemotherapy, such as eribulin mesylate and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic complete response rate (pCR) at the time of definitive surgery.

SECONDARY OBJECTIVES:

I. Determination of the clinical response rate, as measured by clinical exam and imaging studies prior to initiation of therapy and prior to surgery.

II. Measurement of alpha B-crystalline in tissue obtained before initiation of therapy and at the time of definitive surgery.

III. Stem cell markers (cluster of differentiation [CD]44+, CD24-, CD133, aldehyde dehydrogenase 1 [ALDH1] and evaluation of the NOTCH pathway) in tissue obtained before initiation of therapy and at the time of definitive surgery.

IV. Measurement of proliferation markers (Ki67) before and after treatment in tissue obtained before imitation of therapy and at the time of definitive surgery.

V. Measurement of beta III tubulin in tissue obtained before initiation of therapy and at the time of definitive surgery.

VI. Measurement of Tau in tissue obtained before initiation of therapy and at the time of definitive surgery.

VII. Safety evaluation, including following of patients for alopecia and neuropathy.

VIII. Epidermal growth factor receptor (EGFR) staining before and after treatment in tissue obtained before initiation of therapy and at the time of definitive surgery.

OUTLINE:

Patients receive eribulin mesylate intravenously (IV) over 2-5 minutes and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed breast cancer; diagnosis must be reviewed and confirmed by the pathology department at Northwestern Memorial Hospital prior to registration on study, and all biopsy materials need to be reviewed and available for correlative studies
* Patients must have stage I-III breast cancer
* Patients must have estrogen receptor-negative (ER-), progesterone receptor-negative (PR-), human epidermal growth factor receptor 2-negative (Her2-) (0, 1+) or fluorescent in situ hybridization (FISH) < ratio of 1.8
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) by mammogram, ultrasound or physical exam
* Prior diagnosis of cancer is allowed as long as patient is free of disease and has been off treatment for the prior malignancy for a minimal interval of one year
* Patients must have a life expectancy of > 12 weeks
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine transaminase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine: within normal institutional limits
* OR creatinine clearance >= 60 mL/min/1.73^2 for patients with creatinine levels above institutional normal
* Women of childbearing potential must commit to the use of effective contraception while on study
* Eligibility of patients receiving medications of substances known to affect, or with the potential to affect, the activity or pharmacokinetics of eribulin will be determined following review of their use by the Principal Investigator
* All patients must have given signed, informed consent prior to registration on study

Exclusion Criteria:

* Prior chemotherapy, immunotherapy or hormonal therapy for breast cancer is NOT allowed
* Concomitant radiotherapy is NOT allowed
* Patients may NOT be receiving any other investigational agents or concurrent anticancer therapies; in addition, use of any herbal (alternative) medicines is NOT permitted
* Patients with uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations what would limit compliance with study requirements are NOT eligible to participate
* Women who are pregnant or lactating are NOT eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
To determine the pathologic complete response rate (pCR). | Biopsy at baseline and tissue removed at time of surgery (after approximately 12 weeks of neoadjuvant therapy)

SECONDARY OUTCOMES:
Measurement of alpha B-crystalline in tissue obtained | Biopsy at baseline and tissue removed at time of surgery (after approximately 12 weeks of neoadjuvant therapy)
Stem cell markers (CD44+, CD24-, CD133, ALDH1 and evaluation of the NOTCH pathway) in tissue | Biopsy at baseline and tissue removed at time of surgery (after approximately 12 weeks of neoadjuvant therapy)
Measurement of proliferation markers (Ki67) | Biopsy at baseline and tissue removed at time of surgery (after approximately 12 weeks of neoadjuvant therapy)
Measurement of beta III tubulin in tissue | Biopsy at baseline and tissue removed at time of surgery (after approximately 12 weeks of neoadjuvant therapy)
Measurement of Tau in tissue | Biopsy at baseline and tissue removed at time of surgery (after approximately 12 weeks of neoadjuvant therapy)
Determination of the clinical response rate, as measured by clinical exam and imaging studies prior to initiation of therapy and prior to surgery. | Imaging studies at baseline and at time of surgery (after approximately 12 weeks of neoadjuvant therapy)
Safety profile of this drug combination | Symptom assessment prior to each cycle (approximately every 3 weeks) and until resolution 6 months after the last dose of study treatment
EGFR staining before and after treatment | Biopsy at baseline and tissue removed at time of surgery (after approximately 12 weeks of neoadjuvant therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kaklamani, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Kaklamani VG, Jeruss JS, Hughes E, Siziopikou K, Timms KM, Gutin A, Abkevich V, Sangale Z, Solimeno C, Brown KL, Jones J, Hartman AR, Meservey C, Jovanovic B, Helenowski I, Khan SA, Bethke K, Hansen N, Uthe R, Giordano S, Rosen S, Hoskins K, Von Roenn J, Jain S, Parini V, Gradishar W. Phase II neoadjuvant clinical trial of carboplatin and eribulin in women with triple negative early-stage breast cancer (NCT01372579). Breast Cancer Res Treat. 2015 Jun;151(3):629-38. doi: 10.1007/s10549-015-3435-y. Epub 2015 May 26. PMID 26006067